CLINICAL TRIAL: NCT05072522
Title: An Open-label, Multicenter, Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of SKLB1028 in Patients With Advanced Solid Tumors
Brief Title: A Study of SKLB1028 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA114-CSP-012
Record Dates: First submitted 2021-09-26; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — SKLB1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKLB1028 (Experimental): Dose-escalation stage: Patients will receive SKLB1028 capsules orally once daily (QD) in continuous 28-day cycles, in three doses beginning at 200 mg and rising to 400 mg.
  Cohort-expansion stage: Patients will receive SKLB1028 capsules orally once daily (QD) in continuous 28-day cycles at selected dose as per the results of dose-escalation stage.
  Interventions: Drug: SKLB1028

INTERVENTIONS:
Drug: SKLB1028 — SKLB1028 capsules, oral, once daily in continuous 28-day cycles

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of SKLB1028 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is divided into two stages. The first stage is the dose-escalation stage to evaluate the safety, tolerance and pharmacokinetics of SKLB1028 in patients with advanced solid tumors. A classic 3+3 design will be used to determine the maximum tolerated dose (MTD). Patients with advanced solid tumors will receive SKLB1028 orally once daily (QD) in continuous 28-day cycles, starting at a dose of 200 mg and rising to 400 mg. The second stage is cohort-expansion study. The safe tolerated dose group will be selected for case expansion. At this stage, patients with advanced solid tumors with better response on SKLB1028 are mainly enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered to participate in this study and signed the informed consent form.
* Age ≥18, no gender limitation.
* Patients with malignant solid tumor who have failed or could not tolerate standard treatment and for whom no standard treatment is available.
* Recurrent or metastatic solid tumors confirmed by histology; patients who are judged by the investigator to be suitable for treatment with SKLB1028 capsules and who meet the requirements of tumor type for corresponding stages:

  1. Stage I: no restriction on solid tumor types;
  2. Phase II: solid tumor type determined by the investigator and the sponsor based on the results of phase I.
* Stage 1: At least one unmeasurable lesion; Stage 2: At least one measurable lesion according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Patient must meet the following criteria as indicated on the clinical laboratory tests:

  1. Absolute neutrophil count ≥1.5×10^9 /L; platelet count ≥80×10^9 /L; hemoglobin ≥90 g/L;
  2. Serum creatinine ≤ 1.5 × upper limit of normal (ULN);
  3. Total bilirubin ≤ 1.5 × ULN, (≤ 3 × ULN for patients with liver metastasis or liver cancer); Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN (≤ 5 × ULN for patients with liver metastasis or liver cancer).
* Patient is suitable for oral administration of the study drug.
* Female patients should agree to use contraceptive measures (such as IUD, condom, etc.) during the study period and within 6 months after the end of the study; negative serum pregnancy test within 7 days prior to enrollment and must be non-lactating patients; male patients should agree to use contraceptive measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* The patient have a previous history of severe allergy to drugs and food.
* Expected survival < 3 months.
* Other malignant active tumors within the past 3 years; except for cured locally curable cancers, such as basal or squamous cell skin carcinoma, or in situ prostate, cervical or breast cancer.
* Central nervous system metastasis (excluding brain metastasis with stable symptoms after local treatment)
* Patients with hepatitis B (HBsAg positive or HBcAb positive with HBV DNA higher than the upper limit of the normal value of the research center) or hepatitis C (HCV antibody positive with HCV RNA higher than the upper limit of the normal value of the research center) or HIV antibody positive.
* Patients whose toxicity of previous anti-tumor treatment has not recovered to ≤ grade 1.
* Cardiac dysfunction, including:

QTc interval female ≥ 470 ms, male ≥ 450 ms; Complete left bundle branch block, grade II or III atrioventricular block; Poorly controlled malignant arrhythmias; Cardiac valve regurgitation or stenosis requiring treatment; Cardiac ejection fraction less than 50% within 6 months before screening; Myocardial infarction, unstable angina pectoris, severe pericardial disease, severe myocardial disease occurred within 6 months before screening; History of chronic congestive heart failure with NYHA ≥ grade 3.

* Patients have poorly controlled hypertension.
* Patients have thrombotic or embolic events such as cerebrovascular accident, pulmonary embolism, etc within 6 months before screening.
* Patients who have received any antitumor treatment within 4 weeks before the first administration; those who have received herbal or proprietary Chinese medicines with a clear antineoplastic indication 2 weeks prior to the first administration.
* Patients have received other unlisted clinical study drugs within 4 weeks before the first administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  To identify the dose-limited toxicity (DLT).
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 28 days)
  To identify the maximum tolerated dose (MTD）
Treatment Emergent Adverse Event (TEAE) | From the initiation of the first dose to 28 days after the last dose
  TEAE is defined as an adverse event that occurs during treatment

SECONDARY OUTCOMES:
Pharmacokinetic indexes, Cmax | At the end of Cycle 1 (each cycle is 28 days)
  Maximum concentration (Cmax) of SKLB1028
Pharmacokinetic indexes, Tmax Pharmacokinetic indexes, Tmax | At the end of Cycle 1 (each cycle is 28 days)
  Time to Cmax (Tmax) of SKLB1028
Pharmacokinetic indexes, AUC0-t | At the end of Cycle 1 (each cycle is 28 days)
  Area under the concentration-time curve (AUC) from 0 to the last measurable concentration (AUC0-t) of SKLB1028
Overall response rate (ORR) | Up to approximately 2 years
  ORR is defined as the proportion of patients who have a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of first dose until the date of first documented PD as per RECIST 1.1 or death from any cause, whichever occurs first
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of patients who have a response of CR/PR or stable disease (SD) as per RECIST 1.1
Duration of response (DOR) | Up to approximately 2 years
  DoR is defined as the time from the first assessment of CR or PR until the date of first occurrence of progressive disease (PD) as per RECIST 1.1 or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Master, Principal Investigator — Study Principal Investigator
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No